CLINICAL TRIAL: NCT03006666
Title: Integrating Community Health Workers Into Primary Care Teams to Improve Diabetes Prevention in Underserved Communities
Brief Title: Integrating Community Health Workers to Improve Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-00690
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Data Only) (Active Comparator): The teams randomly allocated to the Control Group will not have access to CHWs.
  Interventions: Behavioral: Data Only
- Intervention Group: (CHW Health Coaching Integrated into Team) (Experimental): Teams randomly allocated to the Intervention Group will also receive regular panel data on their pre-DM patients and will have a CHW join the team, attend team meetings, and provide an outreach intervention to all prediabetic patients in the panel, as described below. CHWs and the researchers will provide regular updates to the team on these activities.
  Interventions: Behavioral: CHW Training

INTERVENTIONS:
Behavioral: CHW Training — CHWs will be trained in DM concepts, motivational interviewing, brief action planning, and stages of behavior change. CHWs will participate in a 105- hour core competency training. CHWs will conduct mock telephone counseling calls with trained standardized patients to enhance skills, gain feedback and develop confidence in these techniques.
  In addition to these training experiences, CHWs will have letter templates, motivational interviewing scripts, and protocols available for patient outreach to standardize and guide patient outreach .
  The completion of the CHW training will be followed by a final examination of knowledge and evaluation of trial encounters with "mock" participants (consisting of research staff and advisory board members).
  Individuals who do not pass will receive intensive remediation and be required to repeat the examination.
  Community Health Worker Coaching Intervention.
  Arms: Intervention Group: (CHW Health Coaching Integrated into Team)
Behavioral: Data Only — The teams randomly allocated will not have access to Community Health Workers.
  Arms: Control Group (Data Only)

SUMMARY:
Cluster randomized trial to test the impact of peer health coaches on prediabetic patients. This study will test a scalable model of peer health coaching to address the millions of patients at risk for Diabetes Mellitus, using low cost, culturally congruent personnel to promote prevention of Diabetes Mellitus in patient-centered medical home (PCMH) practice.

DETAILED DESCRIPTION:
This population based trial aims to understand the impact of peer health interventions on panels of patients in a real clinic environment

Investigators will conduct a cluster-randomized trial to test the impact of peer health coaches on prediabetic patients cared for by patient-centered medical home model (PCMH) teams to:

1. Reduce the incidence of type 2 DM in pre-diabetic, PCMH patients;
2. Promote weight loss among pre-diabetic patients;
3. Increase patient activation levels, a measureable construct of engagement, efficacy, skills, and confidence in managing one's health, among pre-DM patients, resulting in:

   1. Improved secondary clinical outcomes: better glycemic and blood pressure control, and lower Framingham risk scores;
   2. Increased utilization of preventive services (e.g. MOVE!, TeleMOVE!, Healthy Lifestyles, etc);
   3. Improved health behaviors (e.g. making dietary and exercise changes); and
4. Develop, implement and assess strategies to recruit, train, and integrate peer CHW health coaches within the PCMH model.

This study will test a scalable model of peer health coaching to address the millions of patients at risk for Diabetes Mellitus (DM),using low cost, culturally congruent personnel to promote prevention of DM in PCMH practice.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one HbA1c result in the prediabetic range (5.7-6.5%) in the 5 years prior to the start date of Phase 2.

Exclusion Criteria:

* A diagnosis of DM, based on ICD-9 codes applied during ambulatory encounters in the 2 years prior to Phase 2
* Treatment with DM medication other than metformin (e.g. insulin or oral agents)
* age greater than 75 years
* exclusion by patient's PCP due to contraindication for lifestyle intervention or CHW outreach.
* Does not speak English or Spanish (necessary to communicate with community health worker)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence rates of type 2 DM | 36 Months
  Cumulative DM incidence rates and time to DM incidence
Weight loss and obesity rates | 36 Months
  Will conduct chi-square test to compare DM incidence rates at 36-months follow-up of the intervention and control arms.
Patient Activation Measure (PAM) scores | 36 Months
  The PAM survey reliably predicts future ER visits, hospital admissions and readmissions, medication adherence and more.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schwartz, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Gupta A, Hu J, Huang S, Diaz L, Gore R, Levy N, Bergman M, Tanner M, Sherman SE, Islam N, Schwartz MD. Implementation fidelity to a behavioral diabetes prevention intervention in two New York City safety net primary care practices. BMC Public Health. 2023 Mar 28;23(1):575. doi: 10.1186/s12889-023-15477-2. PMID 36978071
- [Derived] Islam N, Gepts T, Lief I, Gore R, Levy N, Tanner M, Fang Y, Sherman SE, Schwartz MD. Protocol for the CHORD project (community health outreach to reduce diabetes): a cluster-randomized community health worker trial to prevent diabetes. BMC Public Health. 2018 Apr 19;18(1):521. doi: 10.1186/s12889-018-5419-4. PMID 29673333

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03006666/Prot_SAP_000.pdf